CLINICAL TRIAL: NCT07257250
Title: Effectiveness of Levothyroxine Treatment on In Vitro Fertilization and Pregnancy Outcome in Women With Subclinical Hypothyroidism and Infertility: A Target Trial Emulation
Brief Title: Levothyroxine Treatment and IVF Outcomes in Women With Subclinical Hypothyroidism: A Target Trial Emulation
Acronym: LESI
Status: Recruiting | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 13/25/DD-BVMD
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Subclinical Hypothyroidism; Infertility; Assisted Reproductive Technology; In Vitro Fertilization (IVF); Intracytoplasmic Sperm Injection; Frozen Embryo Transfer (FET)
Keywords: Levothyroxine; Subclinical Hypothyroidism; Infertility; Thyroid Disorders; IVF; ICSI; Frozen Embryo Transfer; FET; Assisted Reproductive Technology; Live Birth; Miscarriage; Pregnancy Outcomes; Thyroid Autoimmunity
MeSH Terms: conditions — Infertility; Thyroid Diseases; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Levothyroxine-Treated Group: Women with subclinical hypothyroidism (TSH 4.2-<10 mIU/L, normal FT4) treated with levothyroxine 25-50 µg/day before frozen embryo transfer (FET). The dose was adjusted every 2-4 weeks to achieve a pre-transfer TSH <2.5 mIU/L. Outcomes including implantation, pregnancy, and live birth rates were assessed after the nearest post-treatment FET cycle.
- Non-Treated (Control) Group: Women with subclinical hypothyroidism (TSH 4.2-<10 mIU/L, normal FT4) who did not receive levothyroxine treatment prior to frozen embryo transfer. Participants were managed expectantly according to clinical judgment. Outcomes were compared with those of the treated group for IVF/ICSI-FET success and pregnancy results.

SUMMARY:
Subclinical hypothyroidism (SCH) is defined by elevated thyroid-stimulating hormone (TSH) with normal free thyroxine (fT4) levels. It affects approximately 5-7% of women of reproductive age and may negatively influence outcomes of assisted reproductive technology (ART). During controlled ovarian stimulation, rising estradiol increases thyroxine-binding globulin and thyroid hormone requirements. These physiological changes, combined with increased metabolic demand in early pregnancy, may worsen SCH and contribute to adverse outcomes such as miscarriage, preterm birth, and hypertensive disorders of pregnancy.

Although levothyroxine (LT4) is routinely used to treat overt hypothyroidism, evidence for its benefit in SCH, especially among infertile women undergoing In Vitro Fertilization (IVF) or Intra-Cytoplasmic Sperm Injection (ICSI) with frozen embryo transfer (FET), remains inconclusive. Some trials and meta-analyses have shown reductions in miscarriage and neonatal mortality, while others have found no improvement in ART or obstetric outcomes.

This study aims to evaluate the effectiveness of levothyroxine therapy on IVF/FET outcomes and subsequent pregnancy results in women with subclinical hypothyroidism and infertility. This retrospective cohort study will emulate the target trial to evaluate whether LT4 treatment, titrated to achieve a pre-transfer TSH < 2.5 mIU/L, improves implantation, live birth, and obstetric outcomes compared with expectant management.

DETAILED DESCRIPTION:
This study is a target trial specified (a randomized controlled trial between the Intervention (Exposed) Group and the Control (Unexposed) Group).

* Intervention (Exposed) Group: Women treated with levothyroxine 25-50 µg/day initiated before the planned FET, titrated every 2-4 weeks to achieve TSH < 2.5 mIU/L before transfer.
* Control (Unexposed) Group: Women managed expectantly without thyroid medication (Before 2020, LT4 use was at the discretion of clinicians; since 2020, the Reproductive Endocrinology Unit has standardized treatment for most SCH patients)

The target trial is emulated using observational data of infertile women aged 18-45 years diagnosed with subclinical hypothyroidism, defined as TSH 4.2-<10 mIU/L and FT4 0.92-1.68 ng/dL, undergoing IVF/ICSI followed by FET in My Duc Hospital and My Duc Phu Nhuan Hospital (Ho Chi Minh City, Vietnam), using routinely collected medical records from January 1, 2019, to December 31, 2024.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years.
* Diagnosed with subclinical hypothyroidism (TSH 4.2-<10 mIU/L with FT4 0.92-1.68 ng/dL).
* Undergoing in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) followed by frozen embryo transfer (FET).

Exclusion Criteria:

* Overt hypothyroidism (TSH ≥10 mIU/L and FT4 ≤0.92 ng/dL).
* Current or recent (within 1 month) use of drugs affecting thyroid function (levothyroxine, amiodarone, methimazole, propylthiouracil).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women aged 18-45 years diagnosed with subclinical hypothyroidism (TSH 4.2-<10 mIU/L, normal FT4) who underwent IVF/ICSI with subsequent frozen embryo transfer (FET) at My Duc Hospital and My Duc Phu Nhuan Hospital, Ho Chi Minh City, Vietnam, between 2019 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after the first frozen embryo transfer (FET) cycle | At delivery (within approximately 9 months after embryo transfer)
  Delivery of a neonate showing any sign of life (heartbeat, umbilical cord pulsation, or movement) at ≥ 22 weeks' gestation after the nearest frozen embryo transfer cycle performed following levothyroxine treatment (or no treatment) in women with subclinical hypothyroidism undergoing IVF/ICSI.

SECONDARY OUTCOMES:
Positive pregnancy test rate | 10-14 days post-transfer
  Serum β-hCG ≥ 25 IU/mL after embryo transfer.
Clinical pregnancy rate | 6 weeks post-transfer
  Ultrasonographic visualization of a gestational sac or embryo with cardiac activity.
Ongoing pregnancy rate | 12 weeks post-transfer
  Presence of a fetus with heartbeat at ≥ 12 weeks' gestation.
Implantation rate | 3 weeks post-transfer
  Number of gestational sacs divided by number of embryos transferred.
Miscarriage rate | Up to 22 weeks post-transfer
  Spontaneous loss of a clinical pregnancy before 22 weeks' gestation.
Ectopic pregnancy rate | Up to 6 weeks post-transfer
  Pregnancy outside the uterine cavity confirmed by ultrasound or surgery.
Multiple pregnancy rate | 6 weeks post-transfer
  Detection of ≥2 gestational sacs on ultrasound.
Preterm birth rate | At delivery
  defined as a birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Gestational hypertension/preeclampsia | After 20 weeks' gestation
  Gestational hypertension/preeclampsia is defined as the development of hypertension with or without proteinuria after 20 weeks of gestation.
Gestational diabetes mellitus | 24-28 weeks' gestation
  Gestational diabetes mellitus is diagnosed by 75-g Oral Glucose Tolerance Test (OGTT) with abnormal fasting or postload glucose at 24-28 weeks.
Neonatal birthweight | At delivery
  Infant weight at delivery (low <2500 g; very low <1500 g; high >4000 g).
Congenital anomalies | at delivery
  Congenital anomalies are defined as structural or functional disorders that occur during intra-uterine life and can be identified prenatally at birth.
Neonatal death | Up to 1 month after delivery
  Death of a live-born infant within 28 days of birth.

CONTACTS AND LOCATIONS:
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poppe K, Glinoer D. Thyroid autoimmunity and hypothyroidism before and during pregnancy. Hum Reprod Update. 2003 Mar-Apr;9(2):149-61. doi: 10.1093/humupd/dmg012. PMID 12751777
- [Background] Zhang Y, Wang H, Pan X, Teng W, Shan Z. Patients with subclinical hypothyroidism before 20 weeks of pregnancy have a higher risk of miscarriage: A systematic review and meta-analysis. PLoS One. 2017 Apr 17;12(4):e0175708. doi: 10.1371/journal.pone.0175708. eCollection 2017. PMID 28414788
- [Background] Bein M, Yu OHY, Grandi SM, Frati FYE, Kandil I, Filion KB. Levothyroxine and the risk of adverse pregnancy outcomes in women with subclinical hypothyroidism: a systematic review and meta-analysis. BMC Endocr Disord. 2021 Feb 27;21(1):34. doi: 10.1186/s12902-021-00699-5. PMID 33639909
- [Background] Maraka S, Singh Ospina NM, O'Keeffe DT, Rodriguez-Gutierrez R, Espinosa De Ycaza AE, Wi CI, Juhn YJ, Coddington CC 3rd, Montori VM, Stan MN. Effects of Levothyroxine Therapy on Pregnancy Outcomes in Women with Subclinical Hypothyroidism. Thyroid. 2016 Jul;26(7):980-6. doi: 10.1089/thy.2016.0014. Epub 2016 May 16. PMID 27112035
- [Background] Kim CH, Ahn JW, Kang SP, Kim SH, Chae HD, Kang BM. Effect of levothyroxine treatment on in vitro fertilization and pregnancy outcome in infertile women with subclinical hypothyroidism undergoing in vitro fertilization/intracytoplasmic sperm injection. Fertil Steril. 2011 Apr;95(5):1650-4. doi: 10.1016/j.fertnstert.2010.12.004. Epub 2010 Dec 30. PMID 21193190
- See also: ClinicalTrials.gov registration (once approved) — https://clinicaltrials.gov/
- See also: University of Medicine and Pharmacy at Ho Chi Minh City - Reproductive Endocrinology Unit — https://ump.edu.vn/